CLINICAL TRIAL: NCT06949150
Title: Combined Coronary CT Angiography and CT Perfusion in Coronary Artery Disease: Integrating Plaque Morphology, Hemodynamics, and Perfusion for Precision Management
Brief Title: Combined Coronary CT Angiography and CT Perfusion in Coronary Artery Disease (CoroFusion)
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-CoroFusion
Record Dates: First submitted 2025-02-09; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-02

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: coronary artery disease, CT angiography, CT perfusion
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Angiography; Nutrition Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conservative group: Patients do not undergo invasive coronary angiography (ICA) and receive medical treatment, lifestyle interventions, or additional tests instead.
  Interventions: Other: Medical therapy
- ICA group: Patients undergo invasive coronary angiography (ICA), with or without percutaneous coronary intervention (PCI), intravascular ultrasound (IVUS), optical coherence tomography (OCT), or fractional flow reserve (FFR).
  Interventions: Diagnostic Test: coronary angiography

INTERVENTIONS:
Diagnostic Test: coronary angiography — Invasive coronary angiography (ICA), with or without percutaneous coronary intervention (PCI), intravascular ultrasound (IVUS), optical coherence tomography (OCT), or fractional flow reserve (FFR).
  Groups: ICA group
Other: Medical therapy — Patients do not undergo invasive coronary angiography (ICA), recieving medical treatment, lifestyle intervention or further test
  Groups: Conservative group

SUMMARY:
Coronary computed tomography angiography (CTA) provides high-resolution imaging of coronary artery disease (CAD), revealing stenosis, plaque characteristics, and hemodynamic markers like CT-derived fractional flow reserve (CT-FFR), axial plaque stress (APS), and wall shear stress (WSS). However, CTA alone has limitations in evaluating the functional significance of lesions, especially in cases with borderline stenosis, severe calcification, or coronary microvascular dysfunction (CMD). CT myocardial perfusion (CTP) complements CTA by directly assessing myocardial blood flow (MBF) and perfusion reserve (MPR), enhancing diagnostic accuracy. Despite its promise, integrating CTA and CTP for comprehensive CAD assessment remains a challenge.

Key gaps include the lack of long-term evidence on combined CTA/CTP findings, particularly in incorporating plaque markers with perfusion deficits. Standardizing ischemic thresholds and validating automated CTP analysis tools remain ongoing challenges. CTP also improves specificity in cases where CTA may overestimate ischemic burden and detects microvascular dysfunction, especially in patients with ischemia and no obstructive CAD (INOCA). Quantitative parameters like MBF have been linked to major adverse cardiovascular events (MACE), but issues with protocol variability and cost-effectiveness persist.

This study, a real-world, single-center observational cohort, evaluates the clinical utility of integrated CTA/CTP imaging in CAD management. It will assess diagnostic synergy, impact on clinical decisions, and prognostic value in predicting 5-year MACE. AI-driven imaging analysis will quantify plaque features and myocardial perfusion defects, integrating multimodal parameters to generate individualized ischemia risk scores. The goal is to refine non-invasive diagnostic pathways and improve CAD management strategies.

DETAILED DESCRIPTION:
Coronary computed tomography angiography (CTA) has transformed the non-invasive assessment of coronary artery disease (CAD) by providing high-resolution visualization of coronary stenosis, plaque characteristics, and emerging hemodynamic parameters such as CT-derived fractional flow reserve (CT-FFR), axial plaque stress (APS), and wall shear stress (WSS). Adverse plaque features, including low-attenuation plaque, napkin-ring sign, positive remodeling, and spotty calcification, have been associated with increased ischemic risk and adverse cardiovascular events. However, CTA alone has inherent limitations in evaluating the functional significance of coronary lesions, particularly in cases of borderline stenosis, diffuse atherosclerosis, severe calcification, and coronary microvascular dysfunction (CMD). CT myocardial perfusion (CTP) serves as a functional complement to CTA by directly assessing myocardial blood flow (MBF), myocardial perfusion reserve (MPR), and time-to-peak (TTP), thereby enhancing diagnostic accuracy and risk stratification in CAD. Despite promising results from previous trials, significant gaps remain in integrating CTA and CTP for comprehensive CAD assessment.

One of the critical gaps is the limited evidence regarding the long-term prognostic implications of combined CTA/CTP findings, particularly when incorporating plaque vulnerability markers (e.g., lipid-rich necrotic core, pericoronary fat attenuation index) with perfusion deficits. Additionally, the quantification of CTP perfusion defects remains an area of active investigation, with ongoing challenges in standardizing ischemic thresholds, optimizing dynamic versus static protocols, and validating automated analysis tools across diverse populations. Furthermore, insufficient data exist on how an integrated anatomical-functional approach influences clinical decision-making, including revascularization strategies, medical therapy optimization, and long-term outcomes in high-risk subgroups such as patients with diabetes, CMD, in-stent restenosis, and severe coronary calcification.

CTP provides unique diagnostic advantages by improving specificity in cases where CTA may overestimate ischemic burden, particularly in moderate stenoses without hemodynamic significance. Moreover, CTP has proven valuable in detecting microvascular dysfunction by identifying impaired MPR in patients with ischemia and no obstructive CAD (INOCA), a population often misclassified by CTA alone. Quantitative perfusion parameters, such as MBF thresholds (<180 mL/100mL/min), have been independently associated with major adverse cardiovascular events (MACE). However, unresolved issues persist, including protocol variability, limited real-world validation of automated perfusion analysis tools, and unclear cost-effectiveness in routine clinical workflows.

This study is a real-world, single-center observational cohort study designed to evaluate the clinical utility of integrated CTA/CTP imaging in CAD management. All treatment decisions will be made jointly by cardiologists and patients based on imaging results and clinical considerations. Patients may undergo medical therapy alone, invasive coronary angiography (ICA) with percutaneous coronary intervention (PCI) when necessary, or additional non-invasive testing such as cardiac magnetic resonance (CMR) or single-photon emission computed tomography (SPECT) for further functional assessment. Our research team will prospectively track the full clinical trajectory of these patients, ensuring comprehensive data collection on diagnostic pathways, therapeutic interventions, and long-term outcomes. At appropriate time points, patients will be stratified into relevant subgroups for detailed analysis.

The primary objectives of this study are threefold: (1) to evaluate the diagnostic synergy of combining CTA-derived stenosis severity, plaque morphology, and hemodynamic markers with CTP-derived ischemic parameters against invasive reference standards such as FFR and coronary flow reserve (CFR); (2) to assess the impact of CTA/CTP-guided strategies on clinical decision-making, including revascularization rates, medical therapy adjustments, and lifestyle interventions; and (3) to determine the prognostic value of combined imaging biomarkers in predicting 5-year MACE, with a focus on sex-specific and diabetes-specific thresholds for ischemia detection.

In addition, this study will perform subgroup analyses to stratify outcomes in high-risk populations, including patients with diabetes and CMD, post-percutaneous coronary intervention (PCI) cohorts with in-stent restenosis or peri-stent plaque progression, and individuals with severe coronary calcification (Agatston score >400), where CTA interpretation remains challenging. Methodologically, the study will incorporate AI-driven imaging analysis for both CTA and CTP. Advanced deep learning algorithms will be used to automatically quantify CTA plaque features, including lipid core volume, fibrous cap thickness, and pericoronary adipose tissue attenuation, improving risk stratification beyond conventional stenosis-based assessments. AI-based CTP analysis will enable automated segmentation and quantification of myocardial perfusion defects, standardizing ischemia thresholds and reducing interobserver variability. Furthermore, machine learning models will integrate multimodal imaging parameters-stenosis severity, plaque vulnerability markers, hemodynamic stress metrics (APS, WSS), and perfusion indices-to generate individualized ischemia risk scores, aiding in personalized treatment decision-making. Advanced hemodynamic modeling using finite element analysis will be employed for CT-FFR and APS computation, validated against invasive pressure wire measurements.

By addressing existing limitations in CAD imaging, this study aims to establish standardized criteria for interpreting combined CTA/CTP findings, provide robust evidence for CTP-guided risk stratification in understudied populations, define the cost-benefit profile of multimodal imaging, and generate a large-scale imaging registry to support future research in precision cardiovascular medicine. The findings from this study are expected to refine non-invasive diagnostic pathways and contribute to the development of personalized, evidence-based strategies for CAD management.

ELIGIBILITY:
Inclusion Criteria:

Patients with an indication for CTP. Qualified patients who have signed a written informed consent form.

Exclusion Criteria:

* Left ventricular ejection fraction < 35%；
* Acute ST-elevation myocardial infarction within 3 months or previous coronary artery bypass graft surgery；
* Planned coronary artery bypass graft surgery after diagnostic angiography；
* Poor quality of CTA/CTP or other reasons by core lab that are unsuitable for plaque, physiological or fat analysis；
* Contraindications for CT perfusion or coronary angiography；
* Coexisting conditions such as pregnancy, cancer, severe valvular heart disease, or liver/kidney dysfunction；
* Other diseases with a life expectancy of less than one year；
* Inability to sign informed consent or, in the researcher's judgment, poor compliance, making it unlikely the patient can complete the study as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for CTP
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | From enrollment to the follow-up of 5 year
  Composite endpoint including cardiovascular death, non-fatal myocardial infarction (MI), hospitalization for unstable angina, and unplanned coronary revascularization.
Diagnostic Accuracy of Combined CTA/CTP vs. Invasive FFR/CFR | 30 days
  Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and area under the ROC curve (AUC) for detecting hemodynamically significant lesions (FFR ≤0.80 or CFR <2.0 or stenosis >90%).
Agreement Between CT-FFR and CTP Perfusion Metrics | 30 days
  Correlation between CT-FFR values and CTP-derived myocardial blood flow (MBF) or perfusion defect size.
Predictive Power of Combined Imaging Biomarkers for MACE | From enrollment to the follow-up of 5 year
  Hazard ratios (HRs) for MACE associated with:High-risk plaque (≥2 adverse features: low-attenuation plaque, positive remodeling, napkin-ring sign, spotty calcification). Perfusion deficit (MBF <150 mL/100mL/min or MPR <1.8). Combined high-risk plaque + perfusion deficit.
Prognostic Utility of Peri-Coronary Fat Attenuation Index (FAI) | From enrollment to the follow-up of 5 year
  Association between elevated FAI (>-70 HU) around stenotic lesions and MACE, adjusted for plaque burden and CTP parameters.

SECONDARY OUTCOMES:
Association Between Perfusion Recovery and Symptom Relief | From enrollment to the follow-up of 1 year
  Percentage of patients with ≥50% reduction in angina episodes linked to normalized MBF (≥200 mL/100mL/min) or MPR (≥2.2) on follow-up CTP.
Dynamic Perfusion Changes in Microvascular Dysfunction | 30 days
  Differences in stress/rest MBF ratios between patients with vs. without coronary microvascular dysfunction (CMD), validated by invasive coronary flow reserve (CFR <2.0).
Sex-Specific Differences in Perfusion-Plaque Relationships | 30 days
  Stratified analysis of plaque-perfusion correlations in women (e.g., higher prevalence of CMD) vs. men.
Impact of Severe Calcification on CTP Diagnostic Accuracy | 30 days
  Sensitivity/specificity of CTP for detecting ischemia in lesions with Agatston score >400, compared to invasive FFR.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No